CLINICAL TRIAL: NCT03502395
Title: Serum Opiorphin Level After Intraoperative Intravenous Lidocaine Infusion and Its Relation to Post-mastectomy Pain: a Prospective Double Blinded Study
Brief Title: Serum Opiorphin Level After Intraoperative Intravenous Lidocaine Infusion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrady S Ibrahim, MD, Assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB0000871246
Record Dates: First submitted 2018-04-11; First posted 2018-04-18 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Cancer, Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Active Comparator): Patients were received intravenous 1 mg/kg of 2 % lidocaine as a loading dose (just before induction of anesthesia) then received 2mg/kg /h lidocaine as maintenance dose (with maximum of 200 mg/h) till the end of the operation (skin closure).
  Interventions: Drug: Lidocaine
- Group II (Placebo Comparator): A standardized equal volume of intravenous bolus dose of normal saline was given as loading dose then normal saline was administered on an equal rate of infusion.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine — ): Patients were received intravenous 1 mg/kg of 2 % lidocaine as a loading dose (just before induction of anesthesia) then received 2mg/kg /h lidocaine as maintenance dose (with maximum of 200 mg/h) till the end of the operation (skin closure).
  Other Names: Active group
  Arms: Group I
Drug: Normal saline — A standardized equal volume of intravenous bolus dose of normal saline was given as loading dose then normal saline was administered on an equal rate of infusion.
  Other Names: Placebo group
  Arms: Group II

SUMMARY:
A prospective, double blinded and randomized study included women with breast cancer and underwent mastectomy, and randomly allocated into two groups of equal size. Lidocaine group and control group.

DETAILED DESCRIPTION:
Women aged between 18 and 60 years old with breast cancer and underwent mastectomy, ASA I or II were included in the study.

* Group I (lidocaine): Patients were received intravenous 1 mg/kg of 2 % lidocaine as a loading dose (just before induction of anesthesia) then received 2mg/kg /h lidocaine as maintenance dose (with maximum of 200 mg/h) till the end of the operation (skin closure).
* Group II (control):- A standardized equal volume of intravenous bolus dose of normal saline was given as loading dose then normal saline was administered on an equal rate of infusion.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 60 years old with breast cancer and underwent mastectomy, American society of Anesthesiologist I or II

Exclusion Criteria:

* Patients with contralateral breast cancer, metastatic tumor, morbid obesity (BMI> 40), allergy to an amide local anesthetic, or morphine sulphate, heart block, renal, or liver dysfunction, or substance abuse disorder, or chronic opioid use

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with breast cancer and underwent mastectomy
Enrollment: 80 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-01-21 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
Serum Opiorphin level | 24 hours postoperative
  Measuring the opiorphin blood level

SECONDARY OUTCOMES:
Visual analog pain score | 24 hours postoperative
  Measure pain intensity. Graded from 0=no pain to 10=worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrady S Ibrahim, M.D., Principal Investigator — Assiut University faculty of medicine
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rougeot C, Robert F, Menz L, Bisson JF, Messaoudi M. Systemically active human opiorphin is a potent yet non-addictive analgesic without drug tolerance effects. J Physiol Pharmacol. 2010 Aug;61(4):483-90. PMID 20814077